CLINICAL TRIAL: NCT05099913
Title: Short-term and Low-dose Application of Neuromodulators Increases Treatment Efficacy and Minimizes Antidepressant Discontinuation Syndrome in Refractory Functional Dyspepsia
Brief Title: The Role of Neuromodulators in Refractory Functional Dyspepsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Shengliang Chen, professor, chief physician, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJYYXHNK
Record Dates: First submitted 2021-09-23; First posted 2021-10-29 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Dyspepsia; Functional Gastrointestinal Disorders; Antidepressant Discontinuation Syndrome; Antidepressant Drug Adverse Reaction
MeSH Terms: conditions — Dyspepsia; Gastrointestinal Diseases | interventions — flupentixol, melitracen drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2-week group (Experimental): Patients were treated with antidepressants for 10-14 days combined with first-class medication(anti-acid drugs, prokinetics), followed by on demand.
  Interventions: Drug: Deanxit
- 4-week group (Experimental): Patients were treated with antidepressants for 4 weeks combined with first-class medication(anti-acid drugs, prokinetics).
  Interventions: Drug: Deanxit

INTERVENTIONS:
Drug: Deanxit — Central neuromodulators was applied in refractory FD patients for different time
  Other Names: Flupentixol and Melitracen

SUMMARY:
The study was designed to investigate the effect of central neuromodulators on refractory functional dyspepsia

DETAILED DESCRIPTION:
Functional dyspepsia (FD) is a prevalent disease combined with emotional disorders. Antidepressants are beneficial in the treatment of refractory FD, while for the long-term use of antidepressants, it could lead to withdrawal syndrome or other adverse events.

Refractory FD patients were unsatisfied with the regular first-line anti-acid treatment. However, many patients were worried about taking antidiepressants, even though guideline has recommended antidepressant use in FD. In our study, we would use low-dose and short-term antidepressant in refractory FD patients, and investigate whether short-term antidepressants application would improve therapeutic efficacy and minimize antidepressant withdrawal of FD patients.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old;
* education level higher than middle school;
* met the Rome IV criteria for FD; absence of abnormalities on physical examination, laboratory tests (including a routine blood test, blood glucose, and liver function examination), and abdominal imaging and GI endoscopy within 6 months;
* absence of Helicobacter pylori infection;
* signed written informed consent for participation in the study.

Exclusion Criteria:

* evidence of organic digestive diseases;
* diabetes, cancer and other diseases might affect GI function;
* pregnancy, lactation or breastfeeding;
* a history of allergic reaction to any of the drugs used in the study;
* participation in other clinical trials in the previous 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline Leeds Dyspepsia Questionnaire (LDQ) scores at 2 weeks and 4 weeks were obtained to assess the dyspepsia outcomes. | 2 weeks and 4 weeks
  The LDQ scores of 0-4 were classified as very mild dyspepsia, 5-8 as mild dyspepsia, 9-15 as moderate dyspepsia, and >15 as severe or very severe dyspepsia.
Changes from baseline Patient Health Questionaire-9 (PHQ-9) scores at 2 weeks and 4 weeks was obtained to assess the depression contition after treatment. | 2 weeks and 4 weeks
  The PHQ-9 scores of 0-4 were classified as none or minimal depression, 5-9 as mild, 10-14 as moderate, 15-19 as moderately severe, and ≥20 as severe depression.
Changes from baseline Generalized Anxiety Questonaire-7 (GAD-7) scores at 2 weeks and 4 weeks were obtained to assess the anxiety contition after treatment. | 2 weeks and 4 weeks
  The GAD-7 scores of 0-4 were classified as the absence of anxiety, 5-9 as mild, 10-14 as moderate, and ≥15 as severe.

SECONDARY OUTCOMES:
Antidepressants discontinuation syndrome was recorded. | 1 week
  Rate of patients with dicscontinuation symdrome including headache, insomia, or flu-like reactions was obtained after antidepressant withdrawal within 1 week.

CONTACTS AND LOCATIONS:
Locations (1):
- Shengliang Chen, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yu YY, Fang DC, Fan LL, Chang H, Wu ZL, Cao Y, Lan CH. Efficacy and safety of esomeprazole with flupentixol/melitracen in treating gastroesophageal reflux disease patients with emotional disorders. J Gastroenterol Hepatol. 2014 Jun;29(6):1200-6. doi: 10.1111/jgh.12552. PMID 24955450
- [Result] Wang L, Zhong Z, Hu J, Rong X, Liu J, Xiao S, Liu Z. Sertraline plus deanxit to treat patients with depression and anxiety in chronic somatic diseases: a randomized controlled trial. BMC Psychiatry. 2015 Apr 14;15:84. doi: 10.1186/s12888-015-0449-2. PMID 25879863
- [Result] Luo L, Du L, Shen J, Cen M, Dai N. Benefit of small dose antidepressants for functional dyspepsia: Experience from a tertiary center in eastern China. Medicine (Baltimore). 2019 Oct;98(41):e17501. doi: 10.1097/MD.0000000000017501. PMID 31593119
- [Result] Fava GA, Gatti A, Belaise C, Guidi J, Offidani E. Withdrawal Symptoms after Selective Serotonin Reuptake Inhibitor Discontinuation: A Systematic Review. Psychother Psychosom. 2015;84(2):72-81. doi: 10.1159/000370338. Epub 2015 Feb 21. PMID 25721705
- [Result] Fava GA, Cosci F. Understanding and Managing Withdrawal Syndromes After Discontinuation of Antidepressant Drugs. J Clin Psychiatry. 2019 Nov 26;80(6):19com12794. doi: 10.4088/JCP.19com12794. PMID 31774947
- [Derived] Wang QQ, Cheng L, Wu BY, Xu P, Qiu HY, Wang B, Yan XJ, Chen SL. Short-course antidepressant therapy reduces discontinuation syndrome while maintaining treatment efficacy in patients with refractory functional dyspepsia: A randomized controlled trial. Front Psychiatry. 2022 Dec 8;13:1063722. doi: 10.3389/fpsyt.2022.1063722. eCollection 2022. PMID 36569610